CLINICAL TRIAL: NCT03321006
Title: Sensation and Psychiatry: Linking Age-Related Hearing Loss to Late-Life Depression and Cognitive Decline
Brief Title: Treating Hearing Loss to Improve Mood and Cognition in Older Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Bret Rutherford, Associate Professor of Clinical Psychiatry, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7540; R21AG059130 (NIH)
Record Dates: First submitted 2017-10-19; First posted 2017-10-25 (Actual); Results first posted 2021-08-19 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Hearing Loss; Depression
Keywords: Aging; Late Life Depression
MeSH Terms: conditions — Hearing Loss; Depression | interventions — Duloxetine Hydrochloride; Escitalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Antidepressant (AD) + full amplification hearing aids (Active Comparator): Participant will be randomized to active comparator and will receive escitalopram or duloxetine + active hearing aid for 12 weeks.
  Interventions: Device: Phonak Audeo B-R 90 hearing aid device (Active); Drug: Duloxetine or escitalopram
- Antidepressant (AD) + Low amplification (sham) hearing aids (Sham Comparator): Participant will be randomized to sham comparator and will receive escitalopram or duloxetine + sham hearing aid for 12 weeks.
  Interventions: Drug: Duloxetine or escitalopram; Device: Audeo B-R 90 hearing aid device (Sham)

INTERVENTIONS:
Device: Phonak Audeo B-R 90 hearing aid device (Active) — Hearing aids will be the latest Audeo B-R 90 devices manufactured by Phonak. Full amplification hearing aids will have their gain determined by audiometric profile as per standard clinical practice
  Arms: Antidepressant (AD) + full amplification hearing aids
Drug: Duloxetine or escitalopram — We opted to allow two potential medication choices so that study participation could be offered to individuals who had previously taken one medication and either not responded or not tolerated it. After 4 weeks if subjects do not meet remission criteria (HRSD≤10), the dose of study medication will be increased to escitalopram 20mg or duloxetine 60mg for the remaining 8 weeks of the study.
  Other Names: Cymbalta or Lexapro
Device: Audeo B-R 90 hearing aid device (Sham) — Hearing aids will be the latest Audeo B-R 90 devices manufactured by Phonak. Low amplification hearing aids will be programmed to a hearing threshold of 10dB across all frequencies
  Arms: Antidepressant (AD) + Low amplification (sham) hearing aids

SUMMARY:
Age-related hearing loss (ARHL) is the third most common health condition affecting older adults after heart disease and arthritis and is the fifth leading cause of years lived with disability worldwide. Many hearing-impaired older adults avoid or withdraw from social contexts in which background noise will make it difficult to communicate, resulting in social isolation and reduced communication with family and friends.Social isolation and loneliness have been linked to numerous adverse physical and mental health outcomes, including dementia, depression, and mortality, and they may also lead to declining physical activity and the development of the syndrome of frailty. In this project it is hypothesized that untreated ARHL represents a distinct route to developing Late-life Depression (LLD) and that individuals with comorbid ARHL/LLD are unlikely to respond to treatments (i.e., antidepressant medication) that do not treat the underlying hearing problem. Initial studies suggest remediation of hearing loss using hearing aids or cochlear implantation may decrease depressive symptoms acutely and over the course of 6 to 12 months follow-up. However, the clinical significance of these findings is obscured by lack of rigorous control groups, failure to objectively document hearing aid compliance, and enrollment of study populations lacking syndromal depression or even a threshold symptom score.

DETAILED DESCRIPTION:
This study will conduct the first clinical trial possessing these design features 40 individuals will be recruited who are aged ≥60 years, diagnosed with a clinically significant depressive disorder, and have moderate ARHL with impaired speech discrimination. Comprehensive baseline psychiatric, audiometric, neuropsychological, and functional assessment will be performed. Participants then will be randomized to receive antidepressant medication (AD) treatment plus full amplification hearing aids or antidepressant medication plus low amplification hearing aids over a 12-week prospective trial. Data from this study could suggest a novel therapeutic strategy for LLD and thereby mitigate its public health burden, while also contributing to the increased recognition and treatment of ARHL more generally.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 60 years
2. diagnosed with Diagnostic and Statistical Manual (DSM) 5 MDD or Persistent Depressive Disorder
3. have duration of depression ≥6 months
4. have 24-item Hamilton Rating Scale for Depression (HRSD) score ≥ 16
5. have moderate to severe symmetric, bilateral hearing loss (combined PTA of >50dB at 2 and 3 kHz)
6. demonstrate impaired speech discrimination scores (60- 100% on 25 word list testing) in one or both ears
7. no prior history of hearing aid use within the past 6 months
8. English speaking
9. are willing to and capable of providing informed consent and complying with study procedures.

Exclusion Criteria:

1. diagnosis of substance abuse or dependence (excluding Tobacco Use Disorder) within the past 12 months
2. history of psychosis, psychotic disorder, mania, or bipolar disorder
3. diagnosis of probable Alzheimer's Disease, Vascular Dementia, or Parkinson's Disease
4. Mini Mental Status Examination (MMSE) ≤ 24
5. current or recent (within the past 4 weeks) treatment with antidepressants, antipsychotics, or mood stabilizers
6. current suicidal ideation (HRSD suicide item > 2) with risk of imminent self-harm
7. any physical or intellectual disability adversely affecting ability to complete assessments
8. acute, severe, or unstable medical or neurological illness
9. contraindication to hearing aid placement
10. significant retrocochlear pathology or organic brain lesion (e.g., acoustic neuroma) responsible for hearing loss.
11. having contraindication (e.g. metal) or unable to tolerate the scanning procedures

Ages: 60 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bret Rutherford, MD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Antidepressant (AD) + Low Amplification (Sham) Hearing Aids | Antidepressant (AD) + Full Amplification Hearing Aids
Started | 14 | 11
Completed | 12 | 11
Not Completed | 2 | 0
Not completed — Death | 1 | 0
Not completed — Lack of Efficacy | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Antidepressant (AD) + Full Amplification Hearing Aids | Antidepressant (AD) + Low Amplification (Sham) Hearing Aids | Total
Number analyzed (Participants) | 11 | 14 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 11 | 14 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.9 (9.2) | 75 (6.5) | 74.1 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 17
  Male | 4 | 4 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 11 | 11 | 22
  Asian | 0 | 1 | 1
  Black/ AA | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 11 | 14 | 25
Hamilton Rating Scale for Depression [Mean (Standard Deviation); unit: units on a scale] — The patient is rated by a clinician among 24 dimensions (24-item HRSD) with a score on a 3 or 5 point scale. Maximum score is a 74. 0-7 are considered as being normal, 8-16 suggest mild depression, 17-23 moderate depression and scores over 24 are indicative of severe depression.
  units on a scale | 19.9 (4.1) | 18.9 (5.4) | 19.4 (4.8)
Social Adjustment Scale- Self Report [Mean (Standard Deviation); unit: units on a scale] — The SAS-SR contains 54 questions that measure instrumental and expressive role performance over the past 2 weeks. Each question is rated on a 5-point scale. The overall adjustment score is obtained by summing the scores of all the items and dividing by the number of items answered.
  The SAS-R overall score ranges from 0-270, with higher questions indication more impairment.
  units on a scale | 2.5 (0.3) | 2.2 (0.4) | 2.3 (0.4)

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Rating Score for Depression (HRSD)
Description: The patient is rated by a clinician among 24 dimensions (24-item HRSD) with a score on a 3 or 5 point scale. Maximum score is a 74. 0-7 are considered as being normal, 8-16 suggest mild depression, 17-23 moderate depression and scores over 24 are indicative of severe depression.
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Antidepressant (AD) + Low Amplification (Sham) Hearing Aids | Antidepressant (AD) + Full Amplification Hearing Aids
Number analyzed (Participants) | 12 | 11
score on a scale | 12.04 (1.72) | 13.86 (1.67)

2. Secondary Outcome: Clinical Global Impression Severity and Improvement (CGI)
Description: Clinical Global Impression - Severity scale (CGI-S) is a 7-point scale (range 0-7) that requires the clinician to rate the severity of the patient's illness at the time of assessment: range is from 0 (=normal, not at all ill) to 7 (=extremely ill, among the most extremely ill patients worsening)
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Antidepressant (AD) + Low Amplification (Sham) Hearing Aids | Antidepressant (AD) + Full Amplification Hearing Aids
Number analyzed (Participants) | 11 | 11
score on a scale | 3.17 (0.33) | 3.20 (0.33)

3. Secondary Outcome: Social Adjustment Scale Self-Report (SAS-SR) Score
Description: The SAS-SR contains 54 questions that measure instrumental and expressive role performance over the past 2 weeks. Each question is rated on a 5-point scale. The overall adjustment score is obtained by summing the scores of all the items and dividing by the number of items answered.
  The SAS-R overall score ranges from 0-270, with higher questions indication more impairment.
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Antidepressant (AD) + Low Amplification (Sham) Hearing Aids | Antidepressant (AD) + Full Amplification Hearing Aids
Number analyzed (Participants) | 11 | 11
score on a scale | 1.96 (0.12) | 2.10 (0.13)

ADVERSE EVENTS:
Time Frame: Adverse Events, Serious Adverse Events, and All-Cause Mortality were assesed over a period of 12 weeks.
Description: Our definition of an an adverse event and/or serious adverse event and/or all-cause mortality did not differ from the definition of adverse event and/or serious adverse event or all-cause mortality from the clinicaltrials.gov definitions. Adverse Events, Serious Adverse Events and All-Cause Mortality was assesed over a period of 12 weeks.
Arm/Group | Antidepressant (AD) + Low Amplification (Sham) Hearing Aids | Antidepressant (AD) + Full Amplification Hearing Aids
All-Cause Mortality (participants affected / at risk) | 1/14 | 0/11
Serious Adverse Events (participants affected / at risk) | 1/14 | 1/11
Other Adverse Events (participants affected / at risk) | 0/14 | 0/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Antidepressant (AD) + Low Amplification (Sham) Hearing Aids (N=14) | Antidepressant (AD) + Full Amplification Hearing Aids (N=11)
Serious Adverse Event (Cardiac disorders) | 0 (0) | 1 (1) — Patient had cardiac history and was started on Wellbutrin. During study was found to have QTC of 532. The patient later informed study psychiatrist that she had a heart attack, though cardiologist thought was unrelated to the Wellbutrin.
All Cause Mortality (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — A patient with pre-existing cancer had cancer return during the study period. The participant was withdrawn from the study at time of diagnosis. We were later informed that patient passed away 4 months after study enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2020-11-06): https://cdn.clinicaltrials.gov/large-docs/06/NCT03321006/Prot_ICF_001.pdf
  • Statistical Analysis Plan (2021-06-02): https://cdn.clinicaltrials.gov/large-docs/06/NCT03321006/SAP_003.pdf